CLINICAL TRIAL: NCT05703191
Title: The Efficacy and Safety of Nitric Oxide Generator and Delivery System in Pulmonary Hypertension of Newborn: A Non-interventional, Observational, Real-world Study
Brief Title: A Real-world Study of Nitric Oxide Generator and Delivery System
Status: Recruiting | Type: Observational
Sponsor: Novlead Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PAH22-09
Record Dates: First submitted 2023-01-06; First posted 2023-01-27 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Hypertension of Newborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nitric Oxide: Inhaled Nitric Oxide
  Interventions: Device: Nitric Oxide Generator and Delivery System

INTERVENTIONS:
Device: Nitric Oxide Generator and Delivery System — Initial at 20ppm is recommended by guidelines. The concentration is adjusted based on actual condition of subjects.

SUMMARY:
The study is aimed to observe the efficacy and safety of Nitric Oxide Generator and Delivery System in Pulmonary Hypertension of Newborn in real clinical settings.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically considered to benefit from inhaled nitric oxide (iNO) and decided to use Nitric Oxide Generator and Delivery System by clinicians
2. Admitted to the Department of Neonatology at the hospital, gender unlimited
3. Diagnosed as pulmonary hypertension and undergoing/decided to undergo respiratory support
4. Documented Oxygenation index (OI) ≥8 prior to the treatment
5. Signed informed consent by the parent(s) or the legal representative(s) with fully aware of the benefits and risks of this study

Exclusion Criteria:

1. Proven risks of nitric oxide contraindication
2. Undergoing or expected to need a combination of other pulmonary vasodilators, surfactants or extracorporeal membrane oxygenation
3. Other circumstances that investigators believe unsuitable for enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newborns
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Oxygenation Index (OI) | Baseline, Minutes 45
  OI = Mean Airway Pressure (MPAW)×100×Fraction of Inspiration Oxygen (FiO2)/Partial Pressure of Oxygen (PaO2)

SECONDARY OUTCOMES:
Change From Baseline in Oxygenation Index (OI) | Baseline, Hour 24, 2 hours after iNO is discontinued
  OI = MPAW×100×FiO2/PaO2
Change From Baseline in Oxygen Saturation | Baseline, Hour 24, 2 hours after iNO is discontinued
  Oxygen Saturation: Peripheral Capillary Oxygen Saturation (SpO2)
Change From Baseline in Pulmonary Artery Pressure (PAP) | Baseline, Hour 24, 2 hours after iNO is discontinued
  Doppler echocardiography is used to detect the regurgitation velocity, and tricuspid regurgitation V values are derived. PAP = 4 × V2 + 5 mmHg.
Percentage of subjects responding to iNO | Hour 24, 2 hours after iNO is discontinued
  Responding to iNO is defined as a decrease in OI of 25% or more
Ventilation and monitoring parameters of Nitric Oxide Generator and Delivery System during treatment | Minutes 45, Hour 24, 2 hours after iNO is discontinued
  Parameters detected by Nitric Oxide Generator and Delivery System
Adverse events | Baseline up to 24 hours after iNO is discontinued
  Incidence of adverse events=Number of subjects with adverse events/Total number of subjects in treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bin Wang, Principal Investigator — Southern Medical University, China
Locations (1):
- ZhuJiang Hospital of Southern Medical University, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No